CLINICAL TRIAL: NCT01123421
Title: Portable Ultrasonometer for Osteoporosis Assessment: Retrospective Fracture Risk Validation Study, Version #1
Brief Title: Develop and Validate Ultrasonic Device for Osteoporotic Fracture Risk Assessment
Acronym: BUSS03
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: BUSS03; 2R44AG017400 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Osteoporosis; Fracture; Aging
Keywords: osteoporosis; fracture risk; aging; tibia; sonometer; ultrasound; BMD; bone mineral density; DXA; 3D-HRpQT; waveform profiles
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With osteoporotic fracture: Approximately 100 postmenopausal women that have been enrolled in a population-based case-control study that have experienced a clinically-diagnosed fracture of thoracolumbar spine or distal forearm due to minimal or moderate trauma based on review on their inpatient and outpatient medical records will be enrolled.
- Without osteoporotic fracture: Approximately 100 control women will have no history of a prior spine, hip, or wrist fracture.

SUMMARY:
Study to demonstrate that the Bone UltraSonic Scanner (BUSS) can aid in detection of osteoporosis and predict prevalent osteoporotic fractures. Measurements derived from the BUSS parameters will be able to discriminate between postmenopausal women with osteoporotic fractures when compared to matched controls without history of osteoporotic fracture.

DETAILED DESCRIPTION:
One of several studies to develop and clinically validate a novel ultrasonographic device, BUSS, for the assessment of osteoporosis and fracture risk.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with osteoporotic fracture at spine or wrist
* postmenopausal women no history of fracture at spine or wrist

Exclusion Criteria:

* women with a history of metabolic disease
* stroke
* tibia fracture or surgery
* BMI ≥ 35 kg/m2
* Teriparatide use currently or within the past 6 months,
* Any skin issues (open wounds or rashes, and/or skin infections) of the tibial area.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both groups
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Determine whether BUSS testing is equivalent or superior to DXA for fracture risk assessment in postmenopausal women. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Armen Sarvazyan, Ph.D., D.Sc., Principal Investigator — Artann Laboratories, Inc.
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States